CLINICAL TRIAL: NCT05956275
Title: Comparison Between USG-Guided Infiltration Popliteal Artery Capsule Knee Block Versus Adductor Canal Block Application as Postoperative Analgesia in Total Knee Prosthesis Under General Anesthesia: Randomized Clinical Trial
Brief Title: USG-Guided Infiltration Popliteal Artery Capsule Knee Block Versus Adductor Canal Block Application as Postoperative Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Siirt Training and Research Hospital (Other Government)
Collaborators: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, asım erçelik, Spesialist Doctor, Siirt Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIBU-TF-AR-AE-001
Record Dates: First submitted 2023-07-04; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Adductor canal block; Infiltration popliteal artery capsule knee block; Tramadol; Bupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adductor canal block and infiltration popliteal artery capsule knee block (Active Comparator): Adductor canal block and infiltration popliteal artery capsule knee block were performed accompanied by USG, Bupivacaine and 10 mL of 0.9% NaCl were applied in each block application.
  Interventions: Drug: Tramadol; Drug: Morfin
- Control (Sham Comparator): No block performed
  Interventions: Drug: Tramadol; Drug: Morfin

INTERVENTIONS:
Drug: Tramadol — ACB and IPACK were performed in USG-guided adductor canal block and infiltration popliteal artery capsule knee block accompanied by USG, Bupivacaine and 10 mL of 0.9% NaCl were applied in each block application.
Drug: Morfin — No block was applied to the patients in control

SUMMARY:
The purpose was to evaluate the effect of USG-guided adductor canal block and infiltration popliteal artery capsule knee block combination on postoperative analgesia before total knee arthroplasty.

DETAILED DESCRIPTION:
In the present study, the purpose was to evaluate the effect of Ultrasound(USG)-guided adductor canal block(ACB) and infiltration popliteal artery capsule knee block(IPACK) combination on postoperative analgesia before total knee arthroplasty(TKA). A total of 40 patients,who were aged 18-75 with the American Society of Anesthesiologists score(ASA) I-III physical status,and who were scheduled for TKA under general anesthesia,were included in the present study.ACB and IPACK were performed in group A(ACB+IPACK) accompanied by USG, Bupivacaine and 10 mL of 0.9% sodium chloride were applied in each block application.No block was applied to the patients in group B.Patient-controlled analgesia was administered to both groups 30 minutes before the end of the surgery.Tramadol HCL was infused at a concentration of 4mg/ml.A bolus of 20 mg of tramadol hydrochloride was given with a lock-in interval of 30 minutes.Postoperative systolic arterial pressure(SAP),diastolic arterial pressure(DAP),mean arterial pressure(MAP),heart rate(HR),visual analog scale(VAS),analgesic consumption,nausea,vomiting, and patient satisfaction scores were recorded.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-75 years
* who were scheduled for elective total knee arthroplasty in Bolu Abant Izzet Baysal University Training and Research Hospital Orthopaedics and Traumatology Clinics

Exclusion Criteria:

* Patients with hypersensitivity to the drugs to be used in the study or the substances in their composition
* pregnant women
* severe cardiac, pulmonary, hepatic, and renal disease
* a history of chronic opioid use and chronic pain syndrome
* patients who were not suitable for regional anesthesia (bleeding diathesis, infection in the procedure area), and those who could not apply patient controlled anesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
tramadol consumption | 24 hours
  tramadol consumption amounts were 0-1 hours, 1-12 hours, 12-24 hours
using morphine as rescue analgesia | 24 hours
  rescue analgesia was evaluated for 0-1 hour, 1-12 hours, and 12-24, the number of patients who used morphine

CONTACTS AND LOCATIONS:
Overall Officials: Kutay Engin Özturan, Professor, Study Chair — Bolu Abant İzzet Baysal University; Cengiz Işık, Professor, Study Chair — Bolu Abant İzzet Baysal University; Asım İlker İtal, MD, Study Chair — Bolu Abant İzzet Baysal University; Mustafa Türkoğlu, MD, Study Chair — Bolu Abant İzzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study is a thesis that I did and presented two years ago. The raw data has not been backed up after going through statistical analysis.

REFERENCES:
- [Result] Allen HW, Liu SS, Ware PD, Nairn CS, Owens BD. Peripheral nerve blocks improve analgesia after total knee replacement surgery. Anesth Analg. 1998 Jul;87(1):93-7. doi: 10.1097/00000539-199807000-00020. PMID 9661553
- [Result] Ryu J, Saito S, Yamamoto K, Sano S. Factors influencing the postoperative range of motion in total knee arthroplasty. Bull Hosp Jt Dis. 1993 Summer;53(3):35-40. PMID 8012266
- [Result] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Result] Lamplot JD, Wagner ER, Manning DW. Multimodal pain management in total knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Feb;29(2):329-34. doi: 10.1016/j.arth.2013.06.005. Epub 2013 Jul 11. PMID 23850410
- [Result] Chia N, Low TC, Poon KH. Peripheral nerve blocks for lower limb surgery--a choice anaesthetic technique for patients with a recent myocardial infarction? Singapore Med J. 2002 Nov;43(11):583-6. PMID 12680529
- [Result] Gurkan Y, Acar S, Solak M, Toker K. Comparison of nerve stimulation vs. ultrasound-guided lateral sagittal infraclavicular block. Acta Anaesthesiol Scand. 2008 Jul;52(6):851-5. doi: 10.1111/j.1399-6576.2008.01655.x. Epub 2008 May 12. PMID 18477077
- [Result] Li D, Yang Z, Xie X, Zhao J, Kang P. Adductor canal block provides better performance after total knee arthroplasty compared with femoral nerve block: a systematic review and meta-analysis. Int Orthop. 2016 May;40(5):925-33. doi: 10.1007/s00264-015-2998-x. Epub 2015 Oct 10. PMID 26452678
- [Result] Shah NA, Jain NP. Is continuous adductor canal block better than continuous femoral nerve block after total knee arthroplasty? Effect on ambulation ability, early functional recovery and pain control: a randomized controlled trial. J Arthroplasty. 2014 Nov;29(11):2224-9. doi: 10.1016/j.arth.2014.06.010. Epub 2014 Jun 19. PMID 25041873
- [Result] Thobhani S, Scalercio L, Elliott CE, Nossaman BD, Thomas LC, Yuratich D, Bland K, Osteen K, Patterson ME. Novel Regional Techniques for Total Knee Arthroplasty Promote Reduced Hospital Length of Stay: An Analysis of 106 Patients. Ochsner J. 2017 Fall;17(3):233-238. PMID 29026354
- [Result] Li JW, Ma YS, Xiao LK. Postoperative Pain Management in Total Knee Arthroplasty. Orthop Surg. 2019 Oct;11(5):755-761. doi: 10.1111/os.12535. PMID 31663286
- [Result] Zhao J, Davis SP. An integrative review of multimodal pain management on patient recovery after total hip and knee arthroplasty. Int J Nurs Stud. 2019 Oct;98:94-106. doi: 10.1016/j.ijnurstu.2019.06.010. Epub 2019 Jun 28. PMID 31352132
- [Result] Li D, Alqwbani M, Wang Q, Liao R, Yang J, Kang P. Efficacy of Adductor Canal Block Combined With Additional Analgesic Methods for Postoperative Analgesia in Total Knee Arthroplasty: A Prospective, Double-Blind, Randomized Controlled Study. J Arthroplasty. 2020 Dec;35(12):3554-3562. doi: 10.1016/j.arth.2020.06.060. Epub 2020 Jun 24. PMID 32680754
- [Result] Canbek U, Akgun U, Aydogan NH, Kilinc CY, Uysal AI. Continuous adductor canal block following total knee arthroplasty provides a better analgesia compared to single shot: A prospective randomized controlled trial. Acta Orthop Traumatol Turc. 2019 Sep;53(5):334-339. doi: 10.1016/j.aott.2019.04.001. Epub 2019 May 2. PMID 31056404
- [Result] Cullom C, Weed JT. Anesthetic and Analgesic Management for Outpatient Knee Arthroplasty. Curr Pain Headache Rep. 2017 May;21(5):23. doi: 10.1007/s11916-017-0623-y. PMID 28283810
- [Result] Chan E, Howle R, Onwochei D, Desai N. Infiltration between the popliteal artery and the capsule of the knee (IPACK) block in knee surgery: a narrative review. Reg Anesth Pain Med. 2021 Sep;46(9):784-805. doi: 10.1136/rapm-2021-102681. Epub 2021 May 14. PMID 33990439
- [Result] Ochroch J, Qi V, Badiola I, Grosh T, Cai L, Graff V, Nelson C, Israelite C, Elkassabany NM. Analgesic efficacy of adding the IPACK block to a multimodal analgesia protocol for primary total knee arthroplasty. Reg Anesth Pain Med. 2020 Oct;45(10):799-804. doi: 10.1136/rapm-2020-101558. Epub 2020 Aug 31. PMID 32868483
- [Result] Tao Y, Zheng SQ, Xu T, Wang G, Wang Y, Wu AS, Yue Y. Median effective volume of ropivacaine 0.5% for ultrasound-guided adductor canal block. J Int Med Res. 2018 Oct;46(10):4207-4213. doi: 10.1177/0300060518791685. Epub 2018 Aug 20. PMID 30124351
- [Result] Jaeger P, Koscielniak-Nielsen ZJ, Hilsted KL, Fabritius ML, Dahl JB. Adductor Canal Block With 10 mL Versus 30 mL Local Anesthetics and Quadriceps Strength: A Paired, Blinded, Randomized Study in Healthy Volunteers. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):553-8. doi: 10.1097/AAP.0000000000000298. PMID 26237001
- [Result] Kampitak W, Tanavalee A, Ngarmukos S, Tantavisut S. Motor-sparing effect of iPACK (interspace between the popliteal artery and capsule of the posterior knee) block versus tibial nerve block after total knee arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2020 Apr;45(4):267-276. doi: 10.1136/rapm-2019-100895. Epub 2020 Feb 4. PMID 32024676
- [Result] Lund J, Jenstrup MT, Jaeger P, Sorensen AM, Dahl JB. Continuous adductor-canal-blockade for adjuvant post-operative analgesia after major knee surgery: preliminary results. Acta Anaesthesiol Scand. 2011 Jan;55(1):14-9. doi: 10.1111/j.1399-6576.2010.02333.x. Epub 2010 Oct 29. PMID 21039357
- [Result] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Result] Xu Z, Zhang H, Luo J, Zhou A, Zhang J. Preemptive analgesia by using celecoxib combined with tramadol/APAP alleviates post-operative pain of patients undergoing total knee arthroplasty. Phys Sportsmed. 2017 Sep;45(3):316-322. doi: 10.1080/00913847.2017.1325312. Epub 2017 May 17. PMID 28475475
- [Result] DeMik DE, Carender CN, Shamrock AG, Callaghan JJ, Bedard NA. Opioid Use After Total Knee Arthroplasty: Does Tramadol Have Lower Risk Than Traditional Opioids? J Arthroplasty. 2020 Jun;35(6):1558-1562. doi: 10.1016/j.arth.2020.01.055. Epub 2020 Jan 28. PMID 32057601
- [Result] Et T, Korkusuz M, Basaran B, Yarimoglu R, Toprak H, Bilge A, Kumru N, Dedeli I. Comparison of iPACK and periarticular block with adductor block alone after total knee arthroplasty: a randomized clinical trial. J Anesth. 2022 Apr;36(2):276-286. doi: 10.1007/s00540-022-03047-6. Epub 2022 Feb 14. PMID 35157136